CLINICAL TRIAL: NCT01653782
Title: Cost Effectiveness of Early Interventions for Non-specific Low Back Pain: A Randomized Controlled Study Investigating Medical Yoga, Exercise Therapy and Evidence Based Advice
Brief Title: Cost Effectiveness of Medical Yoga Therapy on Low Back Pain
Acronym: MYTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Irene Jensen, Professor, Karolinska Institutet
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 6411023
Record Dates: First submitted 2012-06-28; First posted 2012-07-31 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Low Back Pain
Keywords: LPB; RCT; Intervention study; Cost effectiveness; Yoga; evidence based; advice to stay active; exercise training
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- kUNDALINI YOGA (Experimental): Guided kundalini yoga sessions specific for low back pain for 1 hour, twice a week (120 minutes of instructor-led yoga) for 6 weeks. Cd recording for home practice recommended once per day.A written self care pamphlet "The Back book"
  Interventions: Behavioral: Kundalini yoga
- Self care advice to stay active (Active Comparator): Evidence based advice from caregiver to stay active and exercise
  Interventions: Behavioral: Self care advice
- Exercise (Active Comparator): Guided exercise at a gym focusing on strength training. Twice a week during 6 weeks. A written self care pamphlet "The Back book"
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Kundalini yoga — Guided training twice a week for six weeks. Self instructing cd for home practice
  Arms: kUNDALINI YOGA
Behavioral: Self care advice — Evidence based advice from caregiver about keeping active, exercise and a written self care pamphlet "The Back book"
  Arms: Self care advice to stay active
Behavioral: Exercise — Strength training at a gym supervised by a physical therapist twice a week during 6 weeks. Self training instruction was provided. A written self care pamphlet "The Back book"
  Arms: Exercise

SUMMARY:
This randomized controlled study will evaluate the cost effectiveness of a yoga intervention compared to two evidence based programs; giving advice to stay active and guided exercise sessions. The first active program includes a six week standardized strength training program where the participants are personally instructed by a trained physiotherapist. The second active program is a six week standardized kundalini yoga program with group sessions twice a week lead by an experienced yoga instructor. Both programs consist of two exercise sessions per week and lasts for six weeks. After six weeks the participants are instructed to continue practicing their program twice a week on their own. The hypothesis are that a kundalini yoga program as an early intervention for Low Back Pain (LBP) is more cost effective than the two other interventions studied.

Participants were recruited through the occupational health services and by advertisement in the local press. Study subjects eligible for inclusion were informed of the study either by health care personnel at the occupational health care centers or by a research assistant at the Karolinska Institutet. Subjects were informed that if they were eligible to participate in the study they would be given the opportunity to participate in one of three approaches for treatment of neck and back pain.

DETAILED DESCRIPTION:
The study was a randomized control trial with a 12-month follow-up that compared active early intervention using medical yoga with exercise therapy and self-care advice. The medical yoga intervention was a standardized program based on Kundalini yoga. The group was led by an experienced yoga instructor. The exercise therapy was a standardized strength training program led by a trained physiotherapist. Both medical yoga and exercise interventions were held in groups and included two sessions per week over six weeks. After the sixth week, participants were instructed to continue practicing at least twice a week on their own. In the medical yoga group, the participants received written information and a disk providing additional guidance. In the exercise therapy group, the participants received tailored written information on exercise. The third group, evidence-based self-care advice, was physically examined by experienced back pain experts (an orthopedic specialist and a licensed chiropractor), and received an oral recommendation to stay active and a booklet containing evidenced-based self-care advice.

The participants were randomized to one of these three treatment groups after undergoing the initial examination and receiving the evidence-based information on self-care and staying active. The form of randomization was block randomization using the pre-randomization technique, in which for each participant an opaque envelope was picked, in consecutive order, by an external research assistant who had no contact with the participants. After randomization the back pain specialist met with the participants and gave them background information about the intervention they were being offered. Previous studies [19, 20] have shown that expectations of treatment and response levels differ depending on, whether the treatment is physically or psychologically oriented. Therefore, the two training interventions (yoga and exercise therapies) were both presented as well established training therapies, to improve the level of participation and to equalize the participants' expectations of the treatment and its outcomes. After the assignment of study participants to intervention groups, the statistician who performed the analyses on the intervention outcomes was "blinded". This implies that the statistician while assessing the outcomes of the interventions was not aware of the assigned intervention of participants and therefore, was not influenced in any way by the knowledge of which group was the intervention or the control.

Ethical consideration All three groups received treatments based on ethical grounds. The study was approved by the Regional Ethics Committee (2010/108-31/3) and registered in the clinicaltrials.gov protocol registration system (NCT01653782).

Data collection Participants were recruited through the Occupational Health Services (OHS) and by advertisement in the local media in Sweden's Stockholm County. People of working age with neck/back pain were invited to apply for participation in the study. Then, a screening questionnaire was mailed to those who responded to the invitation to participate in the study. Those who scored 90 points or more, i.e., fulfilling the requirements for a yellow flag, on the Örebro Musculoskeletal Pain Screening Questionnaire (OMPSQ) [25] were invited for further physical examination.

The inclusion criteria were having non-specific low back pain, being with the age range of 18-60, having scored 90 points or more on the OMPSQ screening questionnaire and having a sufficient command of Swedish. The exclusion criteria were pregnancy, comorbidities that could affect the ability to perform exercise, ongoing regular weekly yoga practice or strength training and ongoing sickness absences of eight weeks or more.

ELIGIBILITY:
Inclusion Criteria:

* non- specific low back pain,
* 18-60 years old,
* > 90 points on the OMPSQ screening questionnaire for yellow flags and sufficient understanding of the Swedish language

Exclusion Criteria:

* presence of so called Red flags,
* pregnancy,
* comorbidities affecting the ability to perform the interventions,
* presently on sick leave for > 8 weeks,
* ongoing regular weekly yoga practice or strength training.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene B Jensen, PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Friskis och svettis, Stockholm
  - Institute of medical yoga, Stockholm
  - Karolinska instituet, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bramberg EB, Bergstrom G, Jensen I, Hagberg J, Kwak L. Effects of yoga, strength training and advice on back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2017 Mar 29;18(1):132. doi: 10.1186/s12891-017-1497-1. PMID 28356091
- See also: web page for the research group — http://www.ki.se/imm/iir

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment details: period sept 2010-dec 2011, invited to examination at a University clinic. 1st questionnaire ÖMSPQ to screen for risk level, 2nd extensive questionnaire covering multi aspects of back pain,3rd examination by a back specialist, 4th blinded randomisation to allocate to group, 5th information on allocation and evidence based advice
Pre-assignment Details: exclusion: n 12 due to: below 90 on OMSPQ, comorbidities affecting ability to physical activity, not skilled in Swedish language, sick leave exceeding 2 weeks, "red flags"
Groups:
- Exercise: Guided exercise at a gym focusing on strength training. Twice a week during 6 weeks. A written self care pamphlet
- Self Care Advice to Stay Active: Evidence based advice from caregiver to stay active and exercise
  Self care advice : Evidence based advice from caregiver about keeping active, exercise and a written self care pamphlet
- Medical Yoga: Guided kundalini yoga sessions specific for low back pain for 1 hour, twice a week (120 minutes of intructor-led yoga each week) for 6 weeks. Cd recording for home practice recommended once per day.A written self care pamphlet
Period: Overall Study
Arm/Group | Exercise | Self Care Advice to Stay Active | Medical Yoga
Started | 52 | 55 | 52
Completed | 36 | 37 | 46
Not Completed | 16 | 18 | 6
Not completed — Withdrawal by Subject | 9 | 15 | 4
Not completed — Lost to Follow-up | 7 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Medical Yoga: Guided kundalini yoga sessions specific for low back pain for 2 hours, twice a week for 6 weeks. Cd recording for home practice recommended once per day.A written self care pamphlet
- Total: Total of all reporting groups
Arm/Group | Exercise | Self Care Advice to Stay Active | Medical Yoga | Total
Number analyzed (Participants) | 52 | 55 | 52 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 52 | 55 | 52 | 159
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (9.3) | 43.9 (11.7) | 46.9 (9.6) | 45.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 44 | 37 | 113
  Male | 20 | 11 | 15 | 46
Region of Enrollment [Number; unit: participants]
  Sweden | 52 | 55 | 52 | 159

OUTCOME MEASURES:

1. Primary Outcome: Number of Days on Sick Leave
Description: Sick leave using self-reported data on number of days on sick leave
Time Frame: 12 MONTHS
Population: by a power calculation based on estimates of change in the primary outcome variables from earlier studies
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Medical Yoga: Guided kundalini yoga sessions specific for low back pain for 1 hour, twice a week (120 minutes each week of instructor-led yoga) for 6 weeks. Cd recording for home practice recommended once per day.A written self care pamphlet
Arm/Group | Exercise | Self Care Advice to Stay Active | Medical Yoga
Number analyzed (Participants) | 36 | 37 | 46
Days | 9.5 (22.2) | 9.2 (23.1) | 3.6 (6.3)

2. Secondary Outcome: Cost Effectiveness
Description: Assessments of direct and indirect cost. Further, assessments of performance is used to calculate production losses.
Time Frame: 6 months, 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Serious and Other (Not Including Serious) Adverse Events were not collected/assessed.
Groups:
- Medical Yoga: Guided kundalini yoga sessions specific for low back pain for twice a week for 6 weeks. Cd recording for home practice recommended once per day.A written self care pamphlet
Arm/Group | Exercise | Self Care Advice to Stay Active | Medical Yoga
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Problems in recruiting eligible subject and drop outs especially in the control group resulted in a small number of subjects analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No